CLINICAL TRIAL: NCT06023745
Title: Study IL- 35 Level and Fibronectin Type Ⅲ Domain Containing Protein 5 \ Irsin (FNDC5 rs3480) Gene Variations in Chronic Hepatitis B.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Shimaa Badway Hemdan, lecturer of medical biochemistry, Sohag University
Other Study IDs: Soh-Med-23-04-11PD
Record Dates: First submitted 2023-07-17; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Genotype

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case: 30 patients diagnosed as a clinical disease of CHB according to the diagnostic criteria of CHB based on, HBsAg, HBeAg serostatus ,HBV DNA level, biochemical liver function, and ultrasonography
  Interventions: Genetic: genotyping
- control: healthy volunteers with negativity for HBsAg, anti- HCV and anti-HIV and with no abnormalities based on physical examination
  Interventions: Genetic: genotyping

INTERVENTIONS:
Genetic: genotyping — Genotyping. Measurement of SOD serum level. Measurement of IL-35 serum level.

SUMMARY:
Find a possible association between Fibronectin type Ⅲ domain containing protein 5 \ Irsin (FNDC5 rs3480) gene single nucleotide polymorphism with chronic hepatitis B and the distribution of its alleles, in relation to many clinical parameters of the chronic hepatitis B group.

* Asses the correlation between IL-35 serum level and the risk of chronic hepatitis B.
* Asses the correlation between SOD serum level and the risk of chronic hepatitis B.

DETAILED DESCRIPTION:
Hepatitis B virus (HBV) infection is a serious public health problem worldwide, with approximately 2 billion people having a history of HBV infection and 350 million of them suffering from chronic HBV infection (1).

Although the host factors (such as infection age, gender and immune status), viral and environmental factors are thought to be involved in affecting the development of CHB. The mechanisms underlying the different clinical outcomes of HBV infection have not been fully understood. Studies indicated that host genetic factors play a critical role in the development of HBV infection, especially single nucleotide polymorphisms (SNPs), is regarded to be one of the determinants for this clinical heterogeneity(2,3). Some polymorphisms have been reported to be involved in susceptibility to CHB in disease severity and progression, or disease prognosis (4,5).

Irisin is encoded by the FNDC5 gene, whose expression is controlled by the peroxi- some proliferator activated receptor gamma coactivator 1 alpha (PGC-1α). PGC-1α is a transcriptional co-activator which does not bind directly to DNA. Studies indicated that the estrogen-related receptor alpha (ERRα) could be a factor that plays a role in PGC-1α binding to DNA. ERRα is encoded by the ESRRA gene and is an orphan nuclear receptor, which has two domains. One of them allows the interaction with DNA, and the second one with a ligand. The ERRα structure is similar to that of the estrogen receptor alpha (ERα), but this receptor does not bind to natural estrogens. ERRα interacts with a canonical sequence of the estrogen response elements (ERRE). ERRα and ERα could compete with each other to bind to similar DNA elements. Together, ERRα binds to DNA, in complex with PGC-1α, to regulate the activity of genes such as FNDC5 (6).

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed as a clinical disease of CHB according to the diagnostic criteria of CHB based on, HBsAg, HBeAg serostatus ,HBV DNA level, biochemical liver function, and ultrasonography

Exclusion Criteria:

* The chronic HBV patients on antiviral therapy will be excluded.

Ages: 20 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will be conducted on 50 patients 30 patients diagnosed as a clinical disease of CHB according to the diagnostic criteria of CHB based on, HBsAg, HBeAg serostatus ,HBV DNA level, biochemical liver function, and ultrasonography (15) A control group of 30 healthy volunteers with negativity for HBsAg, anti- HCV and anti-HIV and with no abnormalities based on physical examination
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
genotyping of Fibronectin Type Ⅲ Domain Containing Protein 5 \ Irsin (FNDC5 rs3480) | 2 months
  study gene polymorphism of irsin in chronic hepatitis b patients
measure of il 35 in serum | 2 months
  il 35 level in serum of chronic hepatitis b pTIENTS

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Eskandari E, Metanat M, Pahlevani E, Nakhzari-Khodakheir T. Association between TGFbeta1 polymorphisms and chronic hepatitis B infection in an Iranian population. Rev Soc Bras Med Trop. 2017 May-Jun;50(3):301-308. doi: 10.1590/0037-8682-0266-2016. PMID 28700046
- [Background] Blackburn EH. Telomeres and telomerase: the means to the end (Nobel lecture). Angew Chem Int Ed Engl. 2010 Oct 4;49(41):7405-21. doi: 10.1002/anie.201002387. No abstract available. PMID 20821774
- [Background] Nowinska K, Jablonska K, Ciesielska U, Piotrowska A, Haczkiewicz-Lesniak K, Pawelczyk K, Podhorska-Okolow M, Dziegiel P. Association of Irisin/FNDC5 with ERRalpha and PGC-1alpha Expression in NSCLC. Int J Mol Sci. 2022 Nov 17;23(22):14204. doi: 10.3390/ijms232214204. PMID 36430689